CLINICAL TRIAL: NCT05912400
Title: Evaluating Mitochondrial Dysfunction in Patients With Neurofibromatosis Type 1
Status: Completed | Type: Observational
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: 274877
Record Dates: First submitted 2023-05-31; First posted 2023-06-22 (Actual); Results first posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-03

CONDITIONS: Neurofibromatosis 1
MeSH Terms: conditions — Neurofibromatosis 1 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be collected from patients and controls during routine appointments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NF1 Group: This study will look to enroll 40 to 45 adults over 18 years old diagnosed with NF1.
  Interventions: Diagnostic Test: Blood draw; Other: FACIT-F and Pain Scales
- Control Group: This study will look to enroll 10 to 15 adults over 18 years old without NF1.
  Interventions: Diagnostic Test: Blood draw

INTERVENTIONS:
Diagnostic Test: Blood draw — • An additional 10 mL of blood will then be drawn for mitochondrial testing purposes.
Other: FACIT-F and Pain Scales — • Questionnaires regarding pain and fatigue will be provided for the subject to review and answer.
  Groups: NF1 Group

SUMMARY:
Neurofibromatosis type 1 is a common genetic disease with a broad spectrum of clinical manifestations in multiple organs of the body. This project will study the (dys)function of mitochondria in patients with neurofibromatosis through multiple collections of blood samples from patients and people not afflicted by neurofibromatosis (control group). This study will evaluate how the function of mitochondria changes with time and if medications and supplements can influence the function of the mitochondria. Patients will also answer questions regarding symptoms like fatigue and pain.

DETAILED DESCRIPTION:
Neurofibromatosis type 1 is a common genetic disease with a broad spectrum of clinical manifestations in multiple organs of the body. Some of those symptoms are skin lesions, tumors and cancers, as also pain, and fatigue. In animal models of this disease, dysfunction of mitochondria, a part of the cell which is responsible for energy production, is often described. This project will study the (dys)function of mitochondria in patients with neurofibromatosis through multiple collections of blood samples from patients and people not afflicted by neurofibromatosis (control group). Those blood samples will be used to run tests that analyses the function of the mitochondria and compare the results from the neurofibromatosis group with the control group. As multiple samples from the same patient will be tested in different times, this study will evaluate how the function of mitochondria changes with time and if medications and supplements can influence the function of the mitochondria. Patients will also answer questions regarding symptoms like fatigue and pain. Doing so, the investigator plan to confirm mitochondrial dysfunction in patients, if the degree of dysfunction correlates with symptoms like pain and fatigue, and if supplements and medication like MEK inhibitors that patients with neurofibromatosis type 1 use in a daily basis modulates (for better or worse) a pre-existing mitochondrial dysfunction.

ELIGIBILITY:
NF1 Group:

Inclusion Criteria:

* Diagnosed with NF1

Inclusion Criteria:

* Not the first degree relative (biological parent, sibling, or child) of the NF1 patient who is in the NF1 group

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Patients with NF1 at the UAMS Adult NF1 clinic will be invited to participate in the study during their regular clinic appointments.
  * Spouses, friends, and non-relatives of NF1 patients who come to the UAMS Adult NF1 Clinic will be invited to participate in the control arm of the study at the time of the patient appointment.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2023-07-26 (Actual); Primary Completion 2024-08-23 (Actual); Study Completion 2024-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erika Santos Horta, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas For Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- NF1 Group (Longitudinal Group): This study will look to enroll 40 to 45 adults over 18 years old diagnosed with NF1.
  Participants will have SOC labs and an additional 10 mL of blood drawn for mitochondrial testing purposes at Baseline, Week 14, and Week 28. At these same 3 timepoints, measures of fatigue (FACIT-F QoL) and pain (Numeric Pain Rating QoL) will be provided for the participant to review and answer. A medical history will be taken at Baseline only.
- Control Group (Cross-sectional Group): These participants are assessed only at consent, 10 mL of blood will be drawn for mitochondrial testing purposes. They will not receive fatigue or pain measures. Their medical history will not be taken. They will not receive SOC labs.
  This study will look to enroll 10 to 15 adults over 18 years old without NF1.
Period: Overall Study
Arm/Group | NF1 Group (Longitudinal Group) | Control Group (Cross-sectional Group)
Started | 44 | 11
Completed | 36 | 11
Not Completed | 8 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 6 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- NF1 Group (Longitudinal Group): Participants will have SOC labs and an additional 10 mL of blood drawn for mitochondrial testing purposes at Baseline, Week 14, and Week 28. At these same 3 timepoints, measures of fatigue (FACIT-F QoL) and pain (Numeric Pain Rating QoL) will be provided for the participant to review and answer. A medical history will be taken at Baseline only.
  This study will look to enroll 40 to 45 adults over 18 years old diagnosed with NF1.
- Total: Total of all reporting groups
Arm/Group | NF1 Group (Longitudinal Group) | Control Group (Cross-sectional Group) | Total
Number analyzed (Participants) | 44 | 11 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.55 (15.22) | 47.08 (12.93) | 44.26 (14.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 5 | 36
  Male | 13 | 6 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black of African American | 6 | 0 | 6
  Race: White | 36 | 3 | 39
  Race: Other | 1 | 0 | 1
  Race: Unknown or Not Reported | 1 | 8 | 9
Region of Enrollment [Number; unit: participants]
  United States | 44 | 11 | 55
Oxygen Consumption Rate (OCR) [Mean (Standard Deviation); unit: picomole/minute] — Mitochondrial respiration efficiency of PBMCs is measured here by the oxygen consumption rate (OCR) in picomoles/minute. Population: Not all 44 participants with NF1 had OCR values due to timing issues with the blood samples and use of the Seahorse XF bioanalyzer. There were 24 usable blood samples from 24 participants.
  picomole/minute
    number analyzed (Participants) | 24 | 11 | 35
    (all) | 67.71 (19.13) | 53.70 (24.09) | 63.31 (21.49)
Extracellular Acidification Rate (ECAR) [Mean (Standard Deviation); unit: millipH/minute] — Mitochondrial respiration efficiency of PBMCs is measured here by the extracellular acidification rate (ECAR) in millipH/minute. Population: Not all 44 participants with NF1 had OCR values due to the logistics of getting blood samples in time to use the Seahorse XF bioanalyzer. There were 24 usable blood samples from 24 participants.
  millipH/minute
    number analyzed (Participants) | 24 | 11 | 35
    (all) | 29.67 (9.13) | 19.85 (10.64) | 26.58 (10.54)
The Numeric Pain Rating Scale (NRS-11) Current [Mean (Standard Deviation); unit: score on a scale] — The Numeric Pain Rating Scale (NRS-11) asks respondents to make 3 pain ratings (on a scale from 0 to 10, with higher scores indicating greater pain), corresponding to their current pain, their best pain experienced over 24 hours, and their worst pain experienced over 24 hours.
  This is done in 3 visits spanning 28 weeks (14 weeks plus or minus 2 days between visits).
  This study-specific baseline measure is the measure of current pain for participants with NF1. Population: Control participants were not asked to complete this measure.
  score on a scale
    number analyzed (Participants) | 44 | 0 | 44
    (all) | 2.70 (3.137) |  | 2.70 (3.137)
The Numeric Pain Rating Scale (NRS-11) Best [Mean (Standard Deviation); unit: score on a scale] — The Numeric Pain Rating Scale (NRS-11) asks respondents to make 3 pain ratings(on a scale from 0 to 10, with higher scores indicating greater pain), corresponding to their current pain, their best pain experienced over 24 hours, and their worst pain experienced over 24 hours.
  This is done in 3 visits spanning 28 weeks (14 weeks plus or minus 2 days between visits).
  This study-specific measure is the measure of the best pain experienced over 24 hours for participants with NF1. Population: Control participants were not asked to complete this measure.
  score on a scale
    number analyzed (Participants) | 44 | 0 | 44
    (all) | 1.95 (2.605) |  | 1.95 (2.605)
The Numeric Pain Rating Scale (NRS-11) Worst [Mean (Standard Deviation); unit: score on a scale] — The Numeric Pain Rating Scale (NRS-11) asks respondents to make 3 pain ratings (on a scale from 0 to 10, with higher scores indicating greater pain), corresponding to their current pain, their best pain experienced over 24 hours, and their worst pain experienced over 24 hours.
  This is done in 3 visits spanning 28 weeks (14 weeks plus or minus 2 days between visits).
  This study-specific baseline measure is the measure of worst pain experienced over 24 hours for participants with NF1. Population: Control participants were not asked to complete this measure.
  score on a scale
    number analyzed (Participants) | 44 | 0 | 44
    (all) | 4.77 (3.634) |  | 4.77 (3.634)
Functional Assessment of Chronic Illness Therapy (FACIT-F) - Fatigue [Mean (Standard Deviation); unit: score on a scale] — The NF1 clinical symptom of fatigue is measured with the Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F). Population: The control participants were not asked to complete this measure.
  score on a scale
    number analyzed (Participants) | 44 | 0 | 44
    (all) | 71.9943 (19.64485) |  | 71.9943 (19.64485)
Vitamin D [Mean (Standard Deviation); unit: nanogram/milliliter] — The impact of vitamin D treatment to potentially improve mitochondrial function was assessed in units of nanogram/milliliter. Population: The vitamin D levels for control participants were not measured.
  nanogram/milliliter
    number analyzed (Participants) | 44 | 0 | 44
    (all) | 33.666 (13.8982) |  | 33.666 (13.8982)

OUTCOME MEASURES:

1. Primary Outcome: Mitochondrial Respiration Efficiency (as Measured by OCR).
Description: Mitochondrial respiration efficiency is measured here by the oxygen consumption rate (OCR) which is measured in units of picomoles per minute.
Time Frame: Baseline, Week 14, Week 28
Population: The analysis population was determined by how many OCR values (corresponding to blood samples) we had for each visit. We had 24 values for Visit 1, 40 for Visit 2, and 30 for Visit 3 (24+40+30=94). This had to do with logistics (getting blood samples, using the Seahorse XF Bioanalyzer). For the control group, which only had a single blood draw, there were 11 blood samples.
Measure: Mean (Standard Deviation); unit: picomole/minute
Units Other Than Participants: blood sample
Groups:
- NF1 Group (Longitudinal Group): Participants will have SOC labs and an additional 10 mL of blood drawn for mitochondrial testing purposes (OCR and ECAR) at Baseline, Week 14, and Week 28. At these same 3 timepoints, measures of fatigue (FACIT-F QoL) and pain (Numeric Pain Rating QoL) will be provided for the participant to review and answer. A medical history will be taken at Baseline only (vitamin D levels).
  This study will look to enroll 40 to 45 adults over 18 years old diagnosed with NF1.
- Control Group (Cross-sectional Group): These participants are assessed only at consent, 10 mL of blood will be drawn for mitochondrial testing purposes (OCR and ECAR). They will not receive fatigue (FACIT-F) or pain (NRS-11) measures. Their medical history will not be taken (vitamin D levels). They will not receive SOC labs.
  This study will look to enroll 10 to 15 adults over 18 years old without NF1.
Arm/Group | NF1 Group (Longitudinal Group) | Control Group (Cross-sectional Group)
Number analyzed (Participants) | 40 | 11
Number analyzed (blood sample) | 94 | 11
picomole/minute
  Baseline: number analyzed (Participants) | 24 | 11
  Baseline: number analyzed (blood sample) | 24 | 11
  Baseline | 67.7167 (19.13264) | 53.7000 (24.08510)
  Week 14: number analyzed (Participants) | 40 | 0
  Week 14: number analyzed (blood sample) | 40 | 0
  Week 14 | 73.3358 (22.92499) |
  Week 28: number analyzed (Participants) | 30 | 0
  Week 28: number analyzed (blood sample) | 30 | 0
  Week 28 | 68.5789 (17.76314) |
Statistical Analysis 1: Comparison: NF1 Group (Longitudinal Group); Test type: Other; p < 0.01, Spearman's Rho — Spearman's rho was used to analyze correlation between OCR (Oxygen Consumption Rate) and NRS-11 Current (Numeric Pain Rating Scale for current pain)
Statistical Analysis 2: Comparison: NF1 Group (Longitudinal Group); Test type: Other; p = 0.02, Spearman's Rho; Spearman's rho was used to analyze correlation between OCR (Oxygen Consumption Rate) and NRS-11 Best (Numeric Pain Rating Scale for best pain)
Statistical Analysis 3: Comparison: NF1 Group (Longitudinal Group); Test type: Other; p = 0.03, Spearman's Rho; Spearman's rho was used to analyze correlation between OCR (Oxygen Consumption Rate) and NRS-11 Worst (Numeric Pain Rating Scale for worst pain)
Statistical Analysis 4: Comparison: NF1 Group (Longitudinal Group); Test type: Other; p = 0.88, Spearman's Rho; Correlation: OCR (Oxygen Consumption Rate) and FACIT-F TOI (Functional Assessment of Chronic Illness Therapy - Fatigue, Trial Outcome Index)
Statistical Analysis 5: Comparison: NF1 Group (Longitudinal Group); Test type: Other; p = 0.36, Spearman's Rho; Spearman's rho was used to analyze correlation between OCR (Oxygen Consumption Rate) and vitamin D levels

2. Primary Outcome: Mitochondrial Respiration Efficiency (as Measured by ECAR).
Description: Mitochondrial respiration efficiency is measured here by the extracellular acidification rate (ECAR) which is measured in millipH per minute.
Time Frame: Baseline, Week 14, Week 28
Population: The analysis population was determined by how many ECAR values (corresponding to blood samples) we had for each visit. We had 24 values for Visit 1, 40 for Visit 2, and 30 for Visit 3 (24+40+30=94). This had to do with logistics (getting blood samples, using the Seahorse XF Bioanalyzer).
Measure: Mean (Standard Deviation); unit: millipH/minute
Units Other Than Participants: blood sample
Arm/Group | NF1 Group (Longitudinal Group) | Control Group (Cross-sectional Group)
Number analyzed (Participants) | 40 | 11
Number analyzed (blood sample) | 94 | 11
millipH/minute
  Baseline: number analyzed (Participants) | 24 | 11
  Baseline: number analyzed (blood sample) | 24 | 11
  Baseline | 29.6667 (9.13282) | 19.8500 (10.64305)
  Week 14: number analyzed (Participants) | 40 | 0
  Week 14: number analyzed (blood sample) | 40 | 0
  Week 14 | 32.4583 (11.65965) |
  Week 28: number analyzed (Participants) | 30 | 0
  Week 28: number analyzed (blood sample) | 30 | 0
  Week 28 | 33.0467 (7.87990) |
Statistical Analysis 1: Comparison: NF1 Group (Longitudinal Group); Test type: Other; p = 0.54, Spearman's Rho; Spearman's rho used analyze correlation btwn ECAR (Extracellular Acidification Rate) and NRS-11 Current (Numeric Pain Rating Scale for current pain)
Statistical Analysis 2: Comparison: NF1 Group (Longitudinal Group); Test type: Other; p = 0.36, Spearman's Rho; Spearman's rho used to analyze correlation between ECAR (Extracellular Acidification Rate) and NRS-11 Best (Numeric Pain Rating Scale for best pain)
Statistical Analysis 3: Comparison: NF1 Group (Longitudinal Group); Test type: Other; p = 0.94, Spearman's Rho; Spearman's rho used to analyze correlation between ECAR (Extracellular Acidification Rate) & NRS-11 Worst (Numeric Pain Rating Scale for worst pain)
Statistical Analysis 4: Comparison: NF1 Group (Longitudinal Group); Test type: Other; p = 0.53, Spearman's Rho; Correlation: ECAR (Extracellular Acidification Rate) & FACIT-F TOI (Functional Assessment of Chronic Illness Therapy - Fatigue, Trial Outcome Index)
Statistical Analysis 5: Comparison: NF1 Group (Longitudinal Group); Test type: Other; p = 0.51, Spearman's Rho; Spearman's rho was used to analyze correlation between ECAR (Extracellular Acidification Rate) and vitamin D levels

3. Primary Outcome: Vitamin D Levels
Description: We hypothesize that mitochondrial dysfunction among NF1 patients sensitizes them to therapeutic interventions targeting mitochondria. We will assess the impact of vitamin D treatment to potentially improve mitochondrial function as measured by OCR. Vitamin D is measured in units of nanogram per milliliter.
Time Frame: Baseline
Population: The analysis population was determined by how many vitamin D level values were found in the medical records of participants.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter
Arm/Group | NF1 Group (Longitudinal Group) | Control Group (Cross-sectional Group)
Number analyzed (Participants) | 44 | 0
nanogram/milliliter | 33.665909090909 (13.898183638758) |
Statistical Analysis 1: Comparison: NF1 Group (Longitudinal Group); Test type: Other; p = 0.36, Spearman's Rho; Spearman's rho was used to analyze correlation between OCR (Oxygen Consumption Rate) and vitamin D levels
Statistical Analysis 2: Comparison: NF1 Group (Longitudinal Group); Test type: Other; p = 0.51, Spearman's Rho; Spearman's rho was used to analyze correlation between ECAR (Extracellular Acidification Rate) and vitamin D levels

4. Primary Outcome: Pain (as Measured With NRS-11 for Current Pain Over the Past 24 Hours) of NF1 Patients
Description: The NF1 clinical symptom of pain as measured with The Numeric Pain Rating Scale (NRS-11) for current pain over the past 24 hours (min=0, max=10, higher score = more pain). This is done in 3 visits spanning 28 weeks (14 weeks plus or minus 2 days between visits).
Time Frame: Baseline, Week 14, Week 28
Population: The analysis population was determined by how many participants completed the NRS-11 for each visit. We had 44 values for Visit 1, 39 for Visit 2, and 36 for Visit 3 (44+39+36=119).
Measure: Mean (Standard Deviation); unit: Questionnaire score
Units Other Than Participants: Questionnaire score
Arm/Group | NF1 Group (Longitudinal Group) | Control Group (Cross-sectional Group)
Number analyzed (Participants) | 44 | 0
Number analyzed (Questionnaire score) | 119 | 0
Questionnaire score
  Baseline: number analyzed (Questionnaire score) | 44 | 0
  Baseline | 2.70 (3.137) |
  Week 14: number analyzed (Participants) | 39 | 0
  Week 14: number analyzed (Questionnaire score) | 39 | 0
  Week 14 | 2.05 (3.077) |
  Week 28: number analyzed (Participants) | 36 | 0
  Week 28: number analyzed (Questionnaire score) | 36 | 0
  Week 28 | 1.78 (2.706) |
Statistical Analysis 1: Comparison: NF1 Group (Longitudinal Group); Test type: Other; p < 0.01, Spearman's Rho; Spearman's rho was used to analyze correlation between OCR (Oxygen Consumption Rate) and NRS-11 Current (Numeric Pain Rating Scale for current pain)
Statistical Analysis 2: Comparison: NF1 Group (Longitudinal Group); Test type: Other; p = 0.54, Spearman's Rho; Spearman's rho used analyze correlation between ECAR (Extracellular Acidification Rate) & NRS-11 Current (Numeric Pain Rating Scale for current pain)

5. Primary Outcome: Pain (as Measured With NRS-11 for Best Pain Over the Past 24 Hours) of NF1 Patients
Description: The NF1 clinical symptom of pain as measured with The Numeric Pain Rating Scale (NRS-11) for best pain over the past 24 hours (min=0, max=10, higher score = more pain). This is done in 3 visits spanning 28 weeks (14 weeks plus or minus 2 days between visits).
Time Frame: Baseline, Week 14, Week 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Questionnaire score
Units Other Than Participants: Questionnaire score
Arm/Group | NF1 Group (Longitudinal Group) | Control Group (Cross-sectional Group)
Number analyzed (Participants) | 44 | 0
Number analyzed (Questionnaire score) | 119 | 0
Questionnaire score
  Baseline: number analyzed (Questionnaire score) | 44 | 0
  Baseline | 1.95 (2.605) |
  Week 14: number analyzed (Participants) | 39 | 0
  Week 14: number analyzed (Questionnaire score) | 39 | 0
  Week 14 | 1.41 (2.403) |
  Week 28: number analyzed (Participants) | 36 | 0
  Week 28: number analyzed (Questionnaire score) | 36 | 0
  Week 28 | 1.53 (2.324) |
Statistical Analysis 1: Comparison: NF1 Group (Longitudinal Group); Test type: Other; p = 0.02, Spearman's Rho; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: NF1 Group (Longitudinal Group); Test type: Other; p = 0.36, Spearman's Rho; [statistical method as in outcome 2, analysis 2]

6. Primary Outcome: Pain (as Measured With NRS-11 for Worst Pain Over the Past 24 Hours) of NF1 Patients
Description: The NF1 clinical symptom of pain as measured with The Numeric Pain Rating Scale (NRS-11) for worst pain over the past 24 hours (min=0, max=10, higher score = more pain). This is done in 3 visits spanning 28 weeks (14 weeks plus or minus 2 days between visits).
Time Frame: Baseline, Week 14, Week 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Questionnaire score
Units Other Than Participants: Questionnaire score
Arm/Group | NF1 Group (Longitudinal Group) | Control Group (Cross-sectional Group)
Number analyzed (Participants) | 44 | 0
Number analyzed (Questionnaire score) | 119 | 0
Questionnaire score
  Baseline: number analyzed (Questionnaire score) | 44 | 0
  Baseline | 4.77 (3.634) |
  Week 14: number analyzed (Participants) | 39 | 0
  Week 14: number analyzed (Questionnaire score) | 39 | 0
  Week 14 | 3.38 (3.951) |
  Week 28: number analyzed (Participants) | 36 | 0
  Week 28: number analyzed (Questionnaire score) | 36 | 0
  Week 28 | 2.61 (3.433) |
Statistical Analysis 1: Comparison: NF1 Group (Longitudinal Group); Test type: Other; p = 0.03, Spearman's Rho; [statistical method as in outcome 1, analysis 3]
Statistical Analysis 2: Comparison: NF1 Group (Longitudinal Group); Test type: Other; p = 0.94, Spearman's Rho; [statistical method as in outcome 2, analysis 3]

7. Primary Outcome: Fatigue (as Measured FACIT-F TOI) of NF1 Patients.
Description: The NF1 clinical symptom of fatigue as measured with the Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F). This is done in 3 visits spanning 28 weeks (14 weeks plus or minus 2 days between visits).
  The FACIT-F asks respondents to rate items on a scale from 0 to 4. There are 5 subscales with varying possible ranges (due to varying numbers of items) as follows:
  1. Physical Well-Being Subscale: Range 0-28,
  2. Social/Family Well-Being Subscale: Range 0-28,
  3. Emotional Well-Being Subscale: Range 0-24,
  4. Functional Well-Being Subscale: Range 0-28, and
  5. Fatigue Subscale: Range 0-52. The Trial Outcome Index (TOI) is the total score we chose to analyze. It consists of the sum of the Physical Well-Being Subscale, Functional Well-Being Subscale, and Fatigue Subscale and has a score range of 0-108.
  The higher the score, the better the quality of life.
Time Frame: Baseline, Week 14, Week 28
Population: The analysis population was determined by how many participants completed the FACIT-F for each visit. We had 44 values for Visit 1, 39 for Visit 2, and 36 for Visit 3 (44+39+36=119).
Measure: Mean (Standard Deviation); unit: Questionnaire score
Units Other Than Participants: Questionnaire score
Arm/Group | NF1 Group (Longitudinal Group) | Control Group (Cross-sectional Group)
Number analyzed (Participants) | 44 | 0
Number analyzed (Questionnaire score) | 119 | 0
Questionnaire score
  Baseline: number analyzed (Questionnaire score) | 44 | 0
  Baseline | 71.9943 (19.64485) |
  Week 14: number analyzed (Participants) | 39 | 0
  Week 14: number analyzed (Questionnaire score) | 39 | 0
  Week 14 | 73.1752 (17.31894) |
  Week 28: number analyzed (Participants) | 36 | 0
  Week 28: number analyzed (Questionnaire score) | 36 | 0
  Week 28 | 75.3935 (21.97130) |
Statistical Analysis 1: Comparison: NF1 Group (Longitudinal Group); Test type: Other; p = 0.88, Spearman's Rho; [statistical method as in outcome 1, analysis 4]
Statistical Analysis 2: Comparison: NF1 Group (Longitudinal Group); Test type: Other; p = 0.53, Spearman's Rho; [statistical method as in outcome 2, analysis 4]

ADVERSE EVENTS:
Description: Deaths, serious adverse events, and nonserious adverse events were not assessed for study.
Arm/Group | NF1 Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-18): https://cdn.clinicaltrials.gov/large-docs/00/NCT05912400/Prot_SAP_000.pdf